CLINICAL TRIAL: NCT01007643
Title: The Use of Wii Fit ™ to Increase Compliance With Home Exercises for Treatment of Patellofemoral Syndrome in Adolescent Females
Brief Title: Use of Wii Fit (TM) to Increase Compliance With Home Exercises in Treating Patellofemoral Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment of study participants in alloted time and funding
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2009:115
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2010-06

CONDITIONS: Patellofemoral Syndrome; Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
Keywords: anterior knee pain; adolescents; female; interactive video games; patellofemoral syndrome; treatment; compliance; home exercises
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Patient Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wii Fit (TM) Interactive Video Game (Experimental): Wii Fit (TM) Interactive Video Game
  Interventions: Other: Wii Fit (TM) Interactive Video Game
- Traditional Home Exercise Program (Active Comparator): Traditional Home Exercise Program
  Interventions: Other: Traditional Home Exercise Program

INTERVENTIONS:
Other: Wii Fit (TM) Interactive Video Game — Use of interactive video game exercise program on a daily basis focusing on quadriceps and hamstring flexibility along with VMO strengthening.
  Other Names: Nintendo Wii Fit (TM)
  Arms: Wii Fit (TM) Interactive Video Game
Other: Traditional Home Exercise Program — Completion of daily home exercise program for quadriceps and hamstring flexibility and VMO strengthening.
  Arms: Traditional Home Exercise Program

SUMMARY:
To determine the utility of the Wii Fit TM interactive video game program in patellofemoral symptom resolution, development of increased muscle strength and flexibility as a result of increased compliance with home exercises in adolescent females with patellofemoral syndrome.

DETAILED DESCRIPTION:
Patellofemoral syndrome (PFS) is a very common diagnosis amongst adolescents and young adults. Symptoms can be chronic in nature and interfere with sporting activity and activities of daily living. Current treatment consists of home exercises to increase muscular strength and flexibility. Adolescents are known to have poor compliance with treatments for chronic illnesses.

There is a paucity of published literature surrounding the Wii TM Interactive Video Game. There has been one published report of the use of Wii Fit TM in rehabilitation where participants used the Wii Fit TM to train proprioception after ankle injury. Individuals that participated in the Wii Fit TM group found improvement in their balance on objective measures as well as increased enjoyment with their treatment plan. One anecdotal report used the Wii TM video game in physiotherapy treatments of a college athlete and found a dramatic increase in attendance compliance after introduction of the video game.

This randomized controlled study will determine if using the Wii Fit TM for home exercise completion will increase compliance and subsequently improve symptoms related to patellofemoral syndrome in adolescent females.

ELIGIBILITY:
Inclusion Criteria:

* Female between ages of 11 and 17 years of age
* A diagnosis of patellofemoral syndrome with one or more of the following symptoms: anterior knee pain, positive theater sign, stairs provoking knee pain.
* No physiotherapy or regular, structured home exercise program is being followed
* Parental/guardian consent to participate
* Patient assent to participate

Exclusion Criteria:

* Patients participating in physiotherapy at the time of initial assessment or have had physiotherapy in the last 6 months for patellofemoral syndrome
* Patients performing regular home exercise program prescribed by physician, physiotherapist, or other allied health professional for patellofemoral syndrome at time of initial assessment
* Patients who have additional knee pathology (e.g. acute patellar dislocation; acute internal knee derangement (i.e. meniscal, ligament injury); osteochondritis dissecans; severe apophysitis or tendinitis) that could interfere with rehabilitation exercises due to pain or instability from these conditions
* Individuals with history of knee surgery
* Individuals that have a Wii Fit TM video game at home
* Individuals for whom consent and assent is not obtained

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika B Persson, MD, Principal Investigator — University of Manitoba
Locations (1):
- Legacy Sport Medicine, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 females between 11-17 yrs. of age with untreated patellofemoral syndrome recruited from a pediatric sport medicine clinic from October 2009 to June 2010.
Groups:
- Wii Fit (TM) Interactive Video Game: Exercise program involved exercises focusing on VMO strength and hamstring and quadriceps stretching utilizing the Wii Fit (TM) Interactive Video Game. Exercises were to be done on a daily basis for 12 weeks and recorded on the provided exercise calendar.
- Traditional Exercise Program: Exercise programs involved exercises focusing on VMO strength and hamstring and quadriceps stretching. Exercises were to be done on a daily basis for 12 weeks and recorded on the provided exercise calendar.
Period: Overall Study
Arm/Group | Wii Fit (TM) Interactive Video Game | Traditional Exercise Program
Started | 8 | 14
Completed | 8 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wii Fit (TM) Interactive Video Game | Traditional Exercise Program | Total
Number analyzed (Participants) | 8 | 14 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 14 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.6 (1.5) | 13.5 (1.5) | 13.2 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 14 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Exercise Days Completed.
Description: Calculated for the 12 week period as daily exercise completion rate as percentage
Time Frame: 3 months
Population: Per Protocol
Measure: Mean (Full Range); unit: percentage of days completed
Arm/Group | Wii Fit (TM) Interactive Video Game | Traditional Exercise Program
Number analyzed (Participants) | 8 | 14
percentage of days completed | 48.3 [15.7 to 72.6] | 62.4 [20.2 to 91.6]

2. Secondary Outcome: Changes in Patellofemoral Symptoms
Time Frame: 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in Hamstring Flexibility
Time Frame: 3 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Quadriceps Flexibility
Time Frame: 3 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Vastus Medialis Oblique Muscle Strength
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Wii Fit (TM) Interactive Video Game | Traditional Exercise Program
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/14
Other Adverse Events (participants affected / at risk) | 0/8 | 0/14

LIMITATIONS AND CAVEATS:
Early termination of the study lead to less than the required number of study subjects enrolled. Thus secondary outcome measures could not be calculated with certainty.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes